CLINICAL TRIAL: NCT02392325
Title: Evaluation of the Clinical and Immune Response Generated by Heterologous Attenuated Dengue Virus Infection
Brief Title: Evaluating the Clinical and Immune Response to Two Dengue Virus Vaccines in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 302
Record Dates: First submitted 2015-03-02; First posted 2015-03-18 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rDEN1Δ30 and rDEN2Δ30-7169 (Experimental): Participants will receive the rDEN1Δ30 vaccine at Day 0. They will receive the rDEN2Δ30-7169 vaccine at Day 270.
  Interventions: Biological: rDEN1Δ30; Biological: rDEN2Δ30-7169
- Placebo and rDEN2Δ30-7169 (Experimental): Participants will receive placebo vaccine at Day 0. They will receive the rDEN2Δ30-7169 vaccine at Day 270.
  Interventions: Biological: Placebo; Biological: rDEN2Δ30-7169

INTERVENTIONS:
Biological: rDEN1Δ30 — Administered subcutaneously in 0.5 mL containing 10^3.0 plaque-forming units (PFU)
  Arms: rDEN1Δ30 and rDEN2Δ30-7169
Biological: Placebo — Administered subcutaneously in 0.5 mL
  Arms: Placebo and rDEN2Δ30-7169
Biological: rDEN2Δ30-7169 — Administered subcutaneously in 0.5 mL containing 10^3.0 PFU

SUMMARY:
Dengue viruses infect millions of people throughout the tropics and subtropics each year. The development of a dengue vaccine is an important health priority. This study will evaluate the immunologic and clinical response to two dengue vaccines, given 9 months apart, in healthy adults with no history of previous flavivirus infection.

DETAILED DESCRIPTION:
Dengue is a mosquito-borne flavivirus. There are 4 types of dengue virus (DENV-1, DENV-2, DENV-3, and DENV-4), each of which can cause mild illness to life-threatening disease. The purpose of this study is to evaluate the immunologic and clinical response to two dengue vaccines (rDEN1Δ30 and rDEN2Δ30-7169), given 9 months apart, in healthy adults with no history of previous flavivirus infection.

Participants will be randomly assigned to receive the rDEN1Δ30 vaccine or a placebo vaccine at Day 0. Additional study visits will occur at Days 4, 6, 8, 10, 12, 14, 16, 21, 28, 56, 90, 180, and 240. At Day 270, all participants will receive the rDEN2Δ30-7169 vaccine. An inpatient (overnight) stay will occur on Days 274 through 284, with participants being discharged on Day 284, if they meet the study criteria. Additional visits will occur at Days 286, 291, 298, 326, 360, and 450. Study visits will include blood collection and a physical examination. Participants will monitor and record their temperature 3 times a day for several days after each vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female between 18 and 50 years of age, inclusive
* Good general health as determined by physical examination, laboratory screening, and review of medical history
* Available for the duration of the study, approximately 26 weeks post-second inoculation
* Willingness to reside in the inpatient unit for 10 days following receipt of rDEN2Δ30-7169
* Willingness to participate in the study as evidenced by signing the informed consent document
* Females Only: Female participants of childbearing potential willing to use effective contraception. Reliable methods of contraception include: hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, intrauterine device, and abstinence (greater than or equal to 6 months since last sexual encounter). All female participants will be considered having child-bearing potential except for those with hysterectomy, tubal ligation, tubal coil (at least 3 months prior to vaccination), or post-menopausal status documented as at least 1 year since last menstrual period.

Exclusion Criteria:

* Females Only: Currently pregnant, as determined by positive beta-human choriogonadotropin (HCG) test, breastfeeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the requirements of the study protocol
* Evidence of recent opiate use based on urine toxicology screen
* Screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC), alanine aminotransferase (ALT), and serum creatinine, as defined in this protocol
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Any significant alcohol or drug abuse in the past 12 months which has caused medical, occupational, or family problems, as indicated by participant history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the last 6 months)
* HIV infection, by screening and confirmatory assays
* Hepatitis C virus (HCV) infection, by screening and confirmatory assays
* Hepatitis B virus (HBV) infection, by Hepatitis B surface antigen (HBsAg) screening
* Any known immunodeficiency syndrome
* Use of anticoagulant medications (use of antiplatelet medication such as aspirin or non-steroidal anti-inflammatory medication is permitted and will not exclude a participant from enrollment)
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 28 days prior to or following vaccination. Immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone equivalent per day for greater than or equal to 14 days
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 28 days following vaccination
* Asplenia
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 28 days following each vaccination
* History or serologic evidence of previous DENV infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis virus, West Nile virus)
* Previous receipt of a flavivirus vaccine (licensed or investigational)
* Anticipated receipt of any investigational agent in the 28 days before or after each vaccination
* Participant has definite plans to travel to a dengue endemic area during the study
* Inability to comply with the inpatient stay following the second DENV infection
* Refusal to allow storage of specimens for future research

Inclusion Criteria for Inoculation with rDEN2Δ30-7169:

* Good general health as determined by physical examination and review of medical history
* Available for the duration of the study, approximately 26 weeks after the second dose
* Willingness to reside in the inpatient unit for 10 days following receipt of rDEN2Δ30-1769
* Willingness to participate in the study as evidenced by signing the informed consent document
* Females Only: Female participants of childbearing potential willing to use effective contraception for the duration of the trial. Reliable methods of contraception include: hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, intrauterine device, and abstinence (greater than or equal to 6 months since last sexual encounter). All female participants will be considered having child-bearing potential except for those with hysterectomy, tubal ligation, tubal coil (at least 3 months prior to vaccination), or post-menopausal status documented as at least 1 year since last menstrual period.

Exclusion Criteria for Inoculation with rDEN2Δ30-7169:

* Anaphylaxis or angioedema following the first dose of vaccine
* Females Only: Currently pregnant, as determined by positive beta-HCG test, breastfeeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the requirements of the study protocol
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Any significant alcohol or drug abuse in the past 12 months which has caused medical, occupational, or family problems, as indicated by participant history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the last 6 months)
* HIV infection, by screening and confirmatory assays
* HCV infection, by screening and confirmatory assays
* HBV infection, by HBsAg screening
* Any known immunodeficiency syndrome
* Use of anticoagulant medications (use of antiplatelet medication such as aspirin or non-steroidal anti-inflammatory medication is permitted and will not exclude a participant from enrollment)
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 42 days prior to or following vaccination. Immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone equivalent per day for greater than or equal to 14 days.
* Asplenia
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 28 days following vaccination
* Anticipated receipt of any other investigational agent in the 28 days before or after vaccination
* Refusal to allow storage of specimens for future research

Other Treatments and Ongoing Exclusion Criteria:

The following criteria will be reviewed on Study Days 28 and 56 following each vaccination. If any become applicable during the study, the participant will not be included in further immunogenicity evaluations, as of the exclusionary visit. The participant will, however, be encouraged to remain in the study for safety evaluations for the duration of the study.

* Use of any investigational drug or investigational vaccine other than the study vaccine during the 28-day period post-vaccination
* Chronic administration (greater than or equal to 14 days) of steroids (defined as prednisone equivalent of greater than or equal to 10 mg per day), immunosuppressants, or other immune-modifying drugs initiated during the 28-day period post-vaccination (topical and nasal steroids are allowed)
* Receipt of a licensed vaccine during the 28-day period post vaccination
* Receipt of immunoglobulins and/or any blood products during the 28-day period post-vaccination
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Measurement of PRNT50 (plaque reduction neutralization titer) to DENV-1, DENV-2, DENV-3, and DENV-4 | Measured through Day 90 post-vaccination
Incidence of solicited adverse events (AEs) following administration of rDEN2Δ30-7169 at Day 270 | Measured through Day 450
Intensity of solicited adverse events (AEs) following administration of rDEN2Δ30-7169 at Day 270 | Measured through Day 450

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research (CIR), Johns Hopkins School of Public Health
Locations (1):
- Center for Immunization Research, Johns Hopkins School of Public Health, Baltimore, Maryland, United States